CLINICAL TRIAL: NCT02355353
Title: Evaluation of Diffusion Weighted Imaging -MRI in Patients With Resectable Liver Metastases From Colorectal Cancer Treated With Fluoropyrimidine-based Chemotherapy as Preoperative Treatment
Brief Title: Evaluation of Diffusion Weighted Imaging -MRI in Patients With Resectable Liver Metastases From Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EORTC-1423
Record Dates: First submitted 2015-01-27; First posted 2015-02-04 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-01

CONDITIONS: Liver Metastases; Colorectal Cancer
Keywords: DWI-MRI; resectable liver metastases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imaging arm (Experimental)
  Interventions: Other: Experimental: imaging arm

INTERVENTIONS:
Other: Experimental: imaging arm — DWI-MRI scans at baseline, at 14 days after first administration of chemotherapy and after up to 6 cycles of chemotherapy

SUMMARY:
The primary objective of this study is to correlate the percentage change in apparent diffusion coefficient (ADC) between baseline and early therapy (at day 14) with tumor regression grade (TRG) measured in the surgical resection specimen.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm imaging trial. Patients with resectable liver metastases from colorectal cancer (CRC) will undergo Diffusion Weighted Imaging- Magnetic Resonance Imaging (DWI-MRI) scans at least at three separate occasions: at baseline, at 14 days (maximum +/- 1 days deviation is acceptable) after first administration of chemotherapy and finally after up to 6 cycles of chemotherapy (one week prior to surgery).

All patients registered in the study may participate to the test-retest analysis. This analysis required a double baseline scans (called test-retest) to be done on two separate occasions, separated from each other by from one hour to one week but both before start of therapy. The repeated scan at baseline (retest) is optional as it will be used only for the test-retest repeatability analysis.

Dedicated in-house developed software will be used to quantify ADC to assess tumor characteristics and response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven CRC with metachronous or synchronous liver metastases considered to be completely upfront resectable.
* Patients with at least one measurable liver lesion (> 2 cm), measured by contrast CT or MRI at baseline. At least one liver metastasis should be clearly identified and provide a high likelihood of successful resection in the later surgery.
* Patients must be 18 years old or older.
* A World Health Organization (WHO) performance status of 0 or 1.
* Previous adjuvant chemotherapy for primary CRC is allowed if completed at least 12 months before inclusion in this study.
* All the following tests should be done within 6 weeks prior to registration:
* Hematological status: neutrophils (ANC) ≥ 1.5x109/L; platelets ≥ 100x109/L; haemoglobin ≥ 9g/dL.
* Serum creatinine ≤ 1.5 times the upper limit of normal (ULN).
* No significant proteinuria (< 2+ proteinuria on urine dipstick or urine protein < 1g/24 hours urine collection).
* Liver function: serum bilirubin ≤ 1.5 x ULN, alkaline phosphatase, aspartate aminotransferase (ASAT) and alanine aminotransferase (ALAT) ≤ 5x ULN.
* No hypercalcemia: ionized calcium ≤1.5 mmol/L.
* Patients with a buffer range from the normal values of +/- 5% for hematology and +/- 10% for biochemistry are acceptable. This will not apply for Renal Function, including Creatinine.
* Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test within 14 days before trial registration.
* Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 6 months after the last study treatment. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 6 months after the last study treatment.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
* Before patient registration, written informed consent must be given according to International Conference on Harmonization of Good Clinical Practice (ICH/GCP), and national/local regulations.

Exclusion Criteria:

* Evidence of extra-hepatic metastasis (of CRC).
* Previous chemotherapy for metastatic disease or surgical treatment (e.g. surgical resection or radiofrequency ablation) for liver metastasis. Previous radiotherapy or embolization treatment on liver is not allowed.
* Major surgical procedure, open biopsy, or significant traumatic injury in liver within 4 weeks prior to registration.
* Other malignancies in the 3 years prior to study entry with the exception of surgically cured carcinoma in situ of the cervix, in situ breast cancer, incidental finding of stage T1a or T1b prostate cancer, and basal/squamous cell carcinoma of the skin.
* Prior (less than 12 months prior to start treatment) or planned concurrent use of anti-angiogenic drugs such as bevacizumab in the back-bone chemotherapy
* Prior (less than 12 months prior to start treatment) or planned concurrent use of anti-Epidermal Growth Factor Receptor (EGFR) monoclonal Antibody (mAb) such as panitumumab or cetuximab in the back-bone chemotherapy
* Regular use of aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs).
* Ongoing bleeding diathesis (e.g. hemoptysis of ≥ 1/2 teaspoon or 2.5 mL), coagulopathy, or need for administration of full-dose anti-coagulant(s).
* Known history of myocardial infarction and/or stroke within 6 months prior to registration and /or New York Heart Association (NYHA) class III and IV congestive heart failure.
* Uncontrolled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg), or history of hypertensive crisis, or hypertensive encephalopathy.
* History or evidence upon physical examination of Central Nervous System (CNS) metastasis.
* Bowel obstruction.
* Known allergy to any excipient of the standard chemotherapy agents
* Known intolerance to atropine or loperamide.
* Gilbert syndrome.
* Treatment with Cytochrome P450 3A4 (CYP3A4) inducers, unless discontinued > 7 days prior to step 2 of registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-09 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of ADC changes | at day 14 relative to baseline
  Percentage of ADC changes at day 14 relative to baseline
Tumor regression grade (TRG) | After surgery, up to 22 weeks from baseline
  Tumor regression grade (TRG) in the surgical resection specimen

SECONDARY OUTCOMES:
Repeatability Coefficient | from test-retest ADC measurements at baseline
  Repeatability Coefficient from test-retest ADC measurements at baseline
Pre-operative (post-treatment) ADC measurement | up to 21 weeks after baseline
  Pre-operative (post-treatment) ADC measurement
Lesion volume | AT baseline, after 9 weeks and after 18 weeks of chemotherapy
  Lesion volume (baseline and, if applicable, after 3 cycles and after 6 cycles) using radiological assessment
Histopathological measurements of tumor tissue cellularity /density, Necrosis, Proliferation (ki-67) | At baseline and up to 22 weeks after baseline
  Histopathological measurements on liver metastases Tumor tissue cellularity/density, Necrosis, Proliferation (ki-67)

CONTACTS AND LOCATIONS:
Overall Officials: Sigrid Stroobants, Principal Investigator — Universitair Ziekenhuis Brussel